CLINICAL TRIAL: NCT05208788
Title: Estimation of Kidney Function Through a Combination of Renal Urinary Biomarkers in Paediatric Renal Transplant Patients - A Multi-centre Prospective Observational Study
Brief Title: Urinary Biomarkers in Paediatric Kidney Transplantation (pKTx)
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Natural and Medical Sciences Institute (NMI) (Unknown); Cooperative European Paediatric Renal Transplant Initiative (CERTAIN) (Unknown)
Responsible Party: Sponsor
Other Study IDs: pKTx/318/2021BO1
Record Dates: First submitted 2021-07-12; First posted 2022-01-26 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Renal Transplantation; Chronic Kidney Insufficiency; Healthy Controls
Keywords: renal transplantation; biomarkers
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Spot urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Renal transplant patients - group 1: Renal transplant patients with stable renal function parameters (mean SCr (or cystatin C) or mean eGFR based on creatinine and / or cystatin C defined as changes ≤ ±15 % for at least three consecutive ambulatory controls).
  Interventions: Diagnostic Test: Biomarker test
- renal transplant patients - group 2: Renal transplant recipients with stable renal function at inclusion, facing a pre-defined event during the course of the study. Pre-defined events are Acute Rejection (AR), viral transplant-associated infection (e.g. BKV), bacterial infection (febrile urinary tract infection (fUTI)), calcineurin-inhibitor (CNI) toxicity, and acute tubular necrosis (ATN).
  Interventions: Diagnostic Test: Biomarker test
- Patients with Chronic Kidney Disease Stage IV and V (CKD IV-V) - group 3: Patients with CKD IV-V (and maintained urine output, without renal replacement therapy and without pre-defined events).
  Interventions: Diagnostic Test: Biomarker test
- Healthy controls: Healthy children serve as control group
  Interventions: Diagnostic Test: Biomarker test

INTERVENTIONS:
Diagnostic Test: Biomarker test — collection of 500µl to 1 ml of a spot urine sample

SUMMARY:
This study aims to test and validate the panel of study urinary biomarker to assess whether (1) reference values differ between paediatric renal transplant patients, patients with chronic kidney disease stage IV and V (CKD IV-V) and children without any disease, (2) characteristic changes in concentration profile may be observed after event-specific injury, (3) differences between paediatric renal transplant patients with AR and other causes of AKI can be detected, and (4) stratification of renal transplant patients to different histological types of AR is possible.

DETAILED DESCRIPTION:
Despite advances in kidney transplantation, acute rejection (AR) is one of the primary risk factors for allograft kidney injury and function deterioration, and may have a significant impact on long-term graft survival, particularly in paediatric renal transplant patients. Against the background of the limited availability of kidney donor organs, the early recognition of AR is of particular interest to improve long-term allograft survival. Renal allograft biopsy remains the current gold standard for the diagnosis of kidney transplant rejection. However, it is an invasive procedure associated with the risk of bleeding, infection of the renal allograft, arterio-venous fistula, introducing sampling error, and a large inter-observer variation. Therefore, urinary biomarkers from minimally invasive compartments would be helpful for the early detection of clinical rejection before graft functional decline occurs. The current standard monitoring of the renal transplant function includes measurements of serum-creatinine (SCr) levels, estimatedglomerular filtration rate (eGFR), and proteinuria. These markers exhibit a lack of sensitivity and specificity and are late indicators for molecular and cellular events following AR. Furthermore, conditions other than AR (viral and bacterial infection, calcineurin nephrotoxicity, acute ischemic injury) resemble similar morphological features within the renal allograft challenging detection and differentiation of the underlying process. Early treatment of AR could lead to diminished histological injury and improved functional outcome. An intensified immunosuppression management represents the main strategy to counteract the uncontrolled attack of the recipient´s immune system against the renal allograft.

Not surprisingly, many attempts have been made to develop new biomarkers to improve the precision and accuracy in detecting AR for optimizing immunosuppression management. Because allograft reactive cells can gain access to the urinary space, urine represents an appropriate biospecimen to investigate allograft injury. The study urinary biomarkers have been partially discovered and characterized in the past for detection of acute kidney injury (AKI), rarely in renal transplant patients.

This study aims to test and validate the panel of study urinary biomarker to assess whether (1) reference values differ between paediatric renal transplant patients, patients with chronic kidney disease stage IV and V (CKD IV-V) and children without any disease, (2) characteristic changes in concentration profile may be observed after event-specific injury, (3) differences between paediatric renal transplant patients with AR and other causes of AKI can be detected, and (4) stratification of renal transplant patients to different histological types of AR is possible.

ELIGIBILITY:
Inclusion Criteria:

i) Group 1 (patients < 18 years of age)- obtaining reference values without any of the pre-defined events

* renal transplant patients with stable renal function parameters (mean SCr (or cystatin C) or mean eGFR based on creatinine and / or cystatin C defined as changes ≤ ±15 % for at least three consecutive ambulatory controls).
* patients with CKD IV-V (and maintained urine output, without renal replacement therapy and without pre-defined events).
* healthy controls.

Study patients from group 1 may be assigned to the group 2 in the following conditions:

ii) Group 2 (patients < 18 years of age)- obtaining biomarker-specific characteristic in the presence of any of the pre-defined events

* renal transplant recipients with living or deceased kidney transplantation.
* patients with CKD IV-V (and maintained urine output without renal replacement therapy).
* healthy controls.

Exclusion Criteria:

i) Healthy controls

* any comorbidity / medication which may have an impact on urinary biomarker profile (e.g. primary kidney or liver disease, metabolic disease, vasculitis or other immunological disease other than the pre-defined events).
* for group 1: presence of any of the pre-defined event. ii) CKD IV-V
* any comorbidity / medication which may have an impact on urinary biomarker profile (e.g. liver disease, metabolic disease, vasculitis or other immunological disease other than the pre-defined events).
* for group 1: presence of any of the pre-defined event. iii) Renal transplant patients for group 1: presence of any of the pre-defined event.
* Primary non-function of the renal transplant organ.
* Blood group (AB0) incompatible.
* Detection of donor specific antibody (DSA) positive (panel-reactive antibodies) at time of enrolment.
* any comorbidity / medication which may have an impact on urinary biomarker profile (e.g. liver disease, metabolic disease, vasculitis or other immunological disease) other than the pre-defined events.
* Presence of other transplanted organs or co-transplanted organs.
* Intention to not use a standard maintenance immunosuppression regimen consisting of calcineurin inhibitor (CNI), antimetabolite (mycophenolate or azathioprine), inhibitor of mechanistic target of rapamycin (mTOR) (Sirolimus / Everolimus) with/without corticosteroids.
* Any condition that, in the opinion of the investigator, would pose risk to the subject's safe participation, or interfere with their ability to comply with the study requirements, or may impact the quality of the interpretation of the data (e.g. detection of malignancy).
* Failure to collect urine samples or incomplete additional CERTAIN dataset (for collecting information about pre-defined events).

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children < 18 years
Sampling Method: Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Change of serum creatinine level [mg/dl] | from Baseline up to 18 months
  Standard surveillance parameter of kidney function / renal allograft
Change of serum urea level [mg/dl] | from Baseline up to 18 months
  Standard surveillance parameter of kidney function / renal allograft
Change of serum Cystatin C level [mg/l] | from Baseline up to 18 months
  Standard surveillance parameter of kidney function / renal allograft
Measurement of urine creatinine level [g/l] | from Baseline up to 18 months
  Standard surveillance parameter of renal function / renal allograft. All urinary study biomarkers (see below) will be correlated to urine creatinine level [ng/mg Creatinine] and compared with standard surveillance parameters of kidney function / renal allograft (see Outcome 1-3).
Change of urine alpha-1-Microglobulin (A1M) | from Baseline up to 18 months
  Urinary study biomarker. The performance (sensitivity, specificity, positive predictive value and negative predictive value) for detection of kidney / graft deterioration will be calculated using receiver operator characteristics (ROC) curves.
Change of urine Aquaporin 2 (AQP2) [ng/ml] | from Baseline up to 18 months
  Urinary study biomarker. The performance (sensitivity, specificity, positive predictive value and negative predictive value) for detection of kidney / graft deterioration will be calculated using receiver operator characteristics (ROC) curves.
Change of urine Caldesmon [ng/ml] | from Baseline up to 18 months
  Urinary study biomarker. The performance (sensitivity, specificity, positive predictive value and negative predictive value) for detection of kidney / graft deterioration will be calculated using receiver operator characteristics (ROC) curves.
Change of urine Clusterin [ng/ml] | from Baseline up to 18 months
  Urinary study biomarker. The performance (sensitivity, specificity, positive predictive value and negative predictive value) for detection of kidney / graft deterioration will be calculated using receiver operator characteristics (ROC) curves.
Change of urine Cystatin C [ng/ml] | from Baseline up to 18 months
  Urinary study biomarker. The performance (sensitivity, specificity, positive predictive value and negative predictive value) for detection of kidney / graft deterioration will be calculated using receiver operator characteristics (ROC) curves.
Change of urine Interleukin 9 (IL-9) [ng/ml] | from Baseline up to 18 months
  Urinary study biomarker. The performance (sensitivity, specificity, positive predictive value and negative predictive value) for detection of kidney / graft deterioration will be calculated using receiver operator characteristics (ROC) curves.
Change of urine Kidney injury molecule 1 (Kim-1) [ng/ml] | from Baseline up to 18 months
  Urinary study biomarker. The performance (sensitivity, specificity, positive predictive value and negative predictive value) for detection of kidney / graft deterioration will be calculated using receiver operator characteristics (ROC) curves.
Change of urine Nephrin [ng/ml] | from Baseline up to 18 months
  Urinary study biomarker. The performance (sensitivity, specificity, positive predictive value and negative predictive value) for detection of kidney / graft deterioration will be calculated using receiver operator characteristics (ROC) curves.
Change of urine Neutrophil gelatinase-associated lipocalin (NGAL) [ng/ml] | from Baseline up to 18 months
  Urinary study biomarker. The performance (sensitivity, specificity, positive predictive value and negative predictive value) for detection of kidney / graft deterioration will be calculated using receiver operator characteristics (ROC) curves.
Change of urine Osteopontin (OPN) [ng/ml] | from Baseline up to 18 months
  Urinary study biomarker. The performance (sensitivity, specificity, positive predictive value and negative predictive value) for detection of kidney / graft deterioration will be calculated using receiver operator characteristics (ROC) curves.
Change of urine P-selectin (SELP) [ng/ml] | from Baseline up to 18 months
  Urinary study biomarker. The performance (sensitivity, specificity, positive predictive value and negative predictive value) for detection of kidney / graft deterioration will be calculated using receiver operator characteristics (ROC) curves.
Change of urine Podocin [ng/ml] | from Baseline up to 18 months
  Urinary study biomarker. The performance (sensitivity, specificity, positive predictive value and negative predictive value) for detection of kidney / graft deterioration will be calculated using receiver operator characteristics (ROC) curves.
Change of urine Retinol-binding protein 4 (RBP4) [ng/ml] | from Baseline up to 18 months
  Urinary study biomarker. The performance (sensitivity, specificity, positive predictive value and negative predictive value) for detection of kidney / graft deterioration will be calculated using receiver operator characteristics (ROC) curves.
Change of urine Smoothelin [ng/ml] | from Baseline up to 18 months
  Urinary study biomarker. The performance (sensitivity, specificity, positive predictive value and negative predictive value) for detection of kidney / graft deterioration will be calculated using receiver operator characteristics (ROC) curves.
Change of urine Synaptopodin [ng/ml] | from Baseline up to 18 months
  Urinary study biomarker. The performance (sensitivity, specificity, positive predictive value and negative predictive value) for detection of kidney / graft deterioration will be calculated using receiver operator characteristics (ROC) curves.
Change of urine tumour necrosis factor alpha (TNF-α) [ng/ml] | from Baseline up to 18 months
  Urinary study biomarker. The performance (sensitivity, specificity, positive predictive value and negative predictive value) for detection of kidney / graft deterioration will be calculated using receiver operator characteristics (ROC) curves.
Change of urine vascular cell adhesion molecule-1 (VCAM-1) | from Baseline up to 18 months
  Urinary study biomarker. The performance (sensitivity, specificity, positive predictive value and negative predictive value) for detection of kidney / graft deterioration will be calculated using receiver operator characteristics (ROC) curves.

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Weitz, PD Dr. med., Principal Investigator — University Children's Hospital Tuebingen
Locations (1):
- University Children's Hospital Tuebingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No